CLINICAL TRIAL: NCT04134325
Title: A Prospective Pilot Study Assessing the Immunomodulatory Effect and Clinical Activity of Programmed Cell Death Protein 1 Inhibition Following CD30 Directed Chimeric Antigen Receptor T Cell Therapy in Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Study of PD-1 Inhibitors After CD30.CAR T Cell Therapy in Relapsed/Refractory Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1852-ATL
Record Dates: First submitted 2019-09-13; First posted 2019-10-22 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Relapsed Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
Keywords: Classic Hodgkin Lymphoma; Relapsed Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Relapsed/Refractory Hodgkin Lymphoma; CD30; cell therapy; CAR-T; modified T cells; PD-1
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Relapse After Prior CD30 CAR-T Therapy (Experimental): Subjects with relapsed/refractory classical Hodgkin lymphoma (r/r cHL) who have previously progressed on anti-PD-1 therapy, have received a CD30 CAR-T cell therapy and have evidence of progression. Subjects will be offered anti-PD-1 therapy (nivolumab or pembrolizumab, at the discretion of treating oncologist), as per standard of care in r/r cHL.
  Interventions: Biological: Nivolumab; Biological: Pembrolizumab
- Arm 2: Relapse with no Prior CD30 CAR-T Therapy (Experimental): Subjects with relapsed/refractory classical Hodgkin lymphoma (r/r cHL) who have previously progressed on anti-PD-1 therapy, have not received a CD30 CAR-T cell therapy and have evidence of progression. Subjects will be offered anti-PD-1 therapy (nivolumab or pembrolizumab, at the discretion of treating oncologist), as per standard of care in r/r cHL.
  Interventions: Biological: Nivolumab; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Nivolumab — Nivolumab administered at 240mg every two weeks or 480 mg every four weeks as per standard of care after treatment with CD30.CAR T cells
  Other Names: Opdivo
Biological: Pembrolizumab — Pembrolizumab administered at 200 mg every three weeks or 400 mg every six weeks as per standard of care after treatment with CD30.CAR T cells
  Other Names: Keytruda

SUMMARY:
LCCC1852-ATL is a prospective 2-arm study designed to determine if chimeric antigen receptor T (CAR-T) cells result in immunomodulation which can be subsequently exploited by programmed cell death protein 1 (PD-1) antibodies to achieve clinical responses in subjects with relapsed/refractory (r/r) classical Hodgkin Lymphoma (cHL).

DETAILED DESCRIPTION:
In this study, investigators will enroll subjects with relapsed/refractory cHL being treated with anti-PD-1 therapy. The study will examine the treatment of relapsed/refractory cHL in this population in , two arms with 10 subjects each: (1) Arm 1: 10 subjects who have previously received anti-PD-1 therapy and experienced progression and more recently received CD30 CAR-T cell therapy and have evidence of progression, and (2) Arm 2 : 10 subjects who have never received CD30 CAR-T therapy and have evidence of progression are initiating treatment with anti-PD1 therapy. In both arms of the study subjects will be offered anti-PD-1 therapy (nivolumab or pembrolizumab, at the discretion of treating oncologist), as per standard of care in r/r cHL

The primary objective of this study is to estimate the objective response rate (ORR) of anti-PD-1 therapy after progression on CD30 CAR-T cell therapy in study Arm 1 subjects within r/r cHL. The secondary objectives will be to measure the change in T-cell receptor clonality during treatment with anti-PD-1 therapy after progression after CD30 CAR-T therapy in these subjects, the change in peripheral blood immunophenotype during treatment with anti-PD-1 therapy after progression on CD30 CAR-T cell therapy and progression free survival (PFS) of anti-PD-1 therapy after progression on CD30 CAR-T cell therapy.

Preliminary data from subjects treated with anti-PD-1 therapy after progression following CD30 CAR-T cell therapy has suggested surprisingly robust clinical responses to anti-PD-1 therapy. Therefore, this study is an important advancement for understanding both immunomodulation after CD30 CAR-T cell therapy, as well as clinical response to anti-PD-1 therapy. This study will serve as a baseline for clinical response and immunomodulation for future clinical trials evaluating the combination of anti-PD-1 therapy and CD30 CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria for Arm 1: Relapse After Prior CD 30 CAR-T Therapy

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Age ≥18 years at the time of consent.
* Subject is planned to start on standard of care anti-PD-1 therapy per community standards of medical care by their treating oncologist.
* Subject has a diagnosis of relapsed/refractory classical Hodgkin lymphoma after at least three lines of prior therapy with clinical progression after either ATLCAR.CD30 and/or ATLCAR.CD30.CCR4. The CAR-T cell product may be either the UNC, Baylor or Tessa product.
* Subjects with prior allogeneic stem cell transplant will be eligible but will be counseled during consent regarding possible increased risk of graft versus host disease with anti-PD-1 therapy after allogeneic stem cell transplant.
* Subjects must have previously been treated with anti-PD-1 therapy (any anti-PD-1 therapy either standard of care or investigational) prior to receiving autologous CAR-T-cell therapy.
* Subject is willing to provide blood samples that are clinically necessary during anti-PD-1 therapy administered per community standards of medical care.

Inclusion Criteria for Arm 2: Relapse with no Prior CD 30 CAR-T Therapy

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Age ≥18 years at the time of consent.
* Subject is planned to start on standard of care anti-PD-1 therapy per community standards of medical care by their treating oncologist.
* Subject has a diagnosis of classical Hodgkin lymphoma.
* Subjects with prior allogeneic stem cell transplant will be eligible but will be counseled during consent regarding possible increased risk of graft versus host disease with anti-PD-1 therapy after allogeneic stem cell transplant.
* Subject is willing to provide blood samples that are clinically necessary during anti-PD-1 therapy administered per community standards of medical care.
* Subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.
* Subject is willing to consent to study-required blood draws.

Exclusion Criteria for Arm 1: Relapse After Prior CD 30 CAR-T Therapy

* Subject has received anti-CD30 CAR-T therapy within the previous 6 weeks.
* Subject has known active infection with HIV, HTLV, HBV, HCV or any active, uncontrolled infection or sepsis.
* Subject has received chemotherapy or anti-PD-1 therapy following CD30 CAR-T cell product administration.
* Subject has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
* Subject is currently using systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent, or other immunosuppressive medications.

Exclusion Criteria for Arm 2: Relapse with no Prior CD 30 CAR-T Therapy

* Subject has received anti-CD30 CAR-T therapy
* Subject is currently using systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent, or other immunosuppressive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2037-07-07 (Estimated)

PRIMARY OUTCOMES:
Objective response, defined as complete response (CR) or partial response (PR) at 12 weeks after initiating anti-PD-1 therapy | 12 weeks
  Response will be determined by the Lymphoma Response to Immunomodulatory Therapy Criteria in order to evaluate the efficacy of anti-PD-1 therapy after progression on CD30 CAR-T cell therapy in relapsed/refractory (r/r) classical Hodgkin Lymphoma (cHL).

SECONDARY OUTCOMES:
Peripheral T-cell receptor frequency per 100,000 clones on Day 1, Day 21, and Day 42 of anti-PD-1 therapy. | 42 days
  To measure the change in peripheral blood T-cell receptor clonality during treatment with anti-PD-1 therapy after progression on CD30 CAR-T cell therapy.
Percent change in peripheral blood T-cell subsets | 42 days
  Percent change in peripheral blood T-cell subsets will be measured by Fluidigm® based mass cytometry from Day 1 of anti-PD-1 therapy to Day 21 and Day 42 of anti-PD-1 therapy.
Progression free survival | From first day of anti-PD-1 therapy to clinical progression or death, up to 15 years
  Progression free survival of anti-PD-1 therapy after progression on CD30 CAR-T cell therapy will be defined as the duration of time from the first day of anti-PD-1 therapy to clinical progression or death as a result of any cause. Response will be determined by the Lymphoma Response to Immunomodulatory Therapy Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — https://unclineberger.org/